CLINICAL TRIAL: NCT04250961
Title: Pamukkale University Medical Faculty
Brief Title: Effects of Showering in 48-72 Hours of Median Sternotomy on Wound Infection, Pain, Comfort and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fadime Gök, Faculty of Health Sciences, Department of Surgical Disease Nursing, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 60116787-020/24129
Record Dates: First submitted 2020-01-24; First posted 2020-01-31 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Surgical Wound Infection
Keywords: cardiac surgery; pain; patient comfort; satisfaction; showering; wound infection
MeSH Terms: conditions — Surgical Wound Infection; Pain; Personal Satisfaction; Wound Infection

STUDY DESIGN:
Intervention Model Description: A Prospective, Randomized Controlled Trial
Who Masked: Participant
Masking Description: All results (wound culture and photographs) were sent to an Infection Control Committee who was masked as to the patient grouping for evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shower Group (Experimental): Patients who had a shower in 48-72 hours after Median Sternotomy
  Interventions: Other: postoperative early shower
- Control Group (Active Comparator): Patients whose sternal incision site was not connected water until remove sutures
  Interventions: Other: postoperative early shower

INTERVENTIONS:
Other: postoperative early shower — The shower group showered in 48-72 hours after median sternotomy with tap water.

SUMMARY:
Time of showering after surgery is still a controversial issue for surgical patients and health professionals. It has been reported that patients should not shower until sutures are removed since traditionally showering is thought to cause infections after surgery. However, not showering after surgery not only has a negative effect on patient comfort but also brings about the risk of infections.

Sternal wound infections after coronary artery bypass graft surgery through median sternotomy are one of the important, life-threatening complications. For this reasons, the investigators researched the advantages and disadvantages of showering for postoperative sternal wound infections, pain due to sternotomy and patient comfort and satisfaction.

DETAILED DESCRIPTION:
Sternal wound infections after coronary artery bypass graft surgery through median sternotomy are one of the important, life-threatening complications increasing length of hospital stay, morbidity and mortality and difficult to treat. In addition to adopting asepsis and antisepsis, meeting hygiene needs, an important nursing intervention, plays a role in prevention of sternal wound infections.

Showering is an important hygiene practice. It has been reported that patients should not shower until sutures are removed since traditionally showering is thought to cause infections after surgery. However, not showering after surgery not only has a negative effect on patient comfort but also brings about the risk of infections. Guidelines for prevention of surgical site infections do not involve recommendations about early showering after surgery or keeping surgical wounds closed and dry for a long time after surgery.

In recent years, it has been reported that keeping postsurgical wounds closed and dry is unnecessary and that showering before removal of sutures is not harmful. There have been studies which reveal showering early after surgery does not increase the risk of infections, even decreases pain and has a positive influence on patient comfort and satisfaction. It is thought that postsurgical showering can quicken wound healing by cleaning sweat, dirt, microorganisms and debris and thus can reduce the risk of infections. However, at present, whether showering before removal of sutures affects wound healing is debatable. Despite presence of studies about effects of postsurgical showering on wound healing, there have not been any studies on the impact of showering after CABG surgery through median sternotomy. Lack of evidence about this issue causes difficulty in relevant nursing practices.

The present study was performed to evaluate effects of showering in 48-72 hours after median sternotomy on sternal wound infections, sternotomy related pain and patient comfort and satisfaction.

MATERIALS AND METHODS Study Design and Setting This is a randomized controlled study carried out to evaluate effects of showering in 48-72 hours after median sternotomy on sternal wound infections, pain due to sternotomy and patient comfort and satisfaction. The study was conducted in the cardiovascular surgery clinic with 30 beds at a university hospital in Aegean region, Turkey, between 21 December 2016 and 30 September 2017.

Inclusion and Exclusion Criteria Inclusion criteria were age of over 18 years, having CABG surgery through median sternotomy, removal of the chest tube, having sutures in place and accepting to participate in the study. Exclusion criteria were having reoperation, removal of the chest tube 72 hours after surgery, developing complications including cardiac tamponade, pleural effusion and pneumonia after surgery and going to another hospital for follow-up.

The sample size was based on a power analysis made with PS Software Version 3.0.43.17 Since there was not a study about effects of showering in the early postoperative period after sternotomy, the power of the study based on the mean effect size (alpha=0.50), the confidence interval (CI) of 95% and the significance level of P < .05 was determined as 80%.18 The sample size was found to be 50 patients, of whom 25 assigned the intervention group (shower group) and other assigned the control group. Taking account of possible losses, a higher number of subjects at the rate of 20% was planned to include in the study. As a result, each group included 30 subjects. However, four patients, of whom one decided not to shower, one developed sternal instability, one died of aspiration pneumonia on the tenth day of surgery and one went to another hospital for follow-up, were excluded from the shower group. Five patients, of whom one had reoperation on the 13th day due to cardiac tamponade, one died of cardiopulmonary arrest on the 14th day and three went to another hospital for postoperative follow-up, were excluded from the control group. The study was completed with 51 patients, of whom 26 were in the shower group and 25 were in the control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years age and older ,
* Having CABG surgery through median sternotomy,
* Removed the chest tube,
* Must be followed up the same hospital
* Accepting to participate in the study

Exclusion Criteria:

* Having reoperation,
* Having the chest tube until 72 hours after surgery,
* Developed complications including cardiac tamponade, pleural effusion and pneumonia after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-24 (Actual)

PRIMARY OUTCOMES:
Sternotomy on Wound Infection | Symptoms of infection determinated 24 hours after surgery, within 48-72 hours after surgery, up to day 7 post surgery, day 14 post surgery and one month after surgery
  The primary outcome measure was the rate of sternal wound infection. Sternal wound infection was defined as the presence of redness and swelling, or the presence of a purulent exudate or a positive bacterial culture.

SECONDARY OUTCOMES:
The secondary outcomes included sternal wound pain score | wound pain score evaluated within 48-72 hours after surgery (before and after showering), up to day 7 post surgery and day 14 post surgery.
  sternal wound pain score evaluated with visual analog scale. It consists of a vertical or horizontal scale on a 10-cm line, with the 0 cm point corresponding to no pain and 10 cm corresponding to the worst pain.

OTHER OUTCOMES:
Other outcome, patients comfort and satisfaction | patients comfort and satisfaction evaluated by the researcher within 48-72 hours after surgery (before and after showering).
  patients comfort and satisfaction evaluated with using a visual analog scale. It consists of a vertical or horizontal scale on a 10-cm line, with the 0 cm point corresponding to worst comfort and satisfaction and 10 cm corresponding to the best comfort and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Demir Korkmaz, RN, PhD, Study Director — ege university, faculty of nursing; Bilgin Emrecan, Study Chair — Pamukkale University Faculty of Medicine
Locations (1):
- Fadime Gök, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gok F, Demir Korkmaz F, Emrecan B. The effects of showering in 48-72 h after coronary artery bypass graft surgery through median sternotomy on wound infection, pain, comfort, and satisfaction: randomized controlled trial. Eur J Cardiovasc Nurs. 2022 Jan 11;21(1):56-66. doi: 10.1093/eurjcn/zvab010. PMID 33871023